CLINICAL TRIAL: NCT02036164
Title: Randomized Controlled Trial Comparing Concurrent Chemoradiation Versus Concurrent Chemoradiation Followed by Adjuvant Chemotherapy in Locally Advanced Cervical Cancer Patients
Brief Title: Adjuvant Chemotherapy for Locally Advanced Cervical Cancer
Acronym: ACT-LACC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Siriwan Tangjitgamol, MD (Other)
Collaborators: National Research Council of Thailand (Other Government); Navamindradhiraj University (Other); Chiang Mai University (Other); Prince of Songkla University (Other); Bhumibol Adulyadej Hospital (Other); Lopburi Cancer Hospital (Unknown); Ubonratchathani Cancer Hospital (Unknown); Udonthani Cancer Hospital (Unknown); Chonburi Cancer Hospital (Unknown); Lampang Cancer Hospital (Other); Health Intervention and Technology Assessment Program (Unknown); Rajburi Hospital (Unknown)
Responsible Party: Sponsor-Investigator, Siriwan Tangjitgamol, MD, Doctor, Navamindradhiraj University
Organization: Navamindradhiraj University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: COA-CREC 002/2013; 20140106001 (Registry Identifier: TCTR)
Record Dates: First submitted 2014-01-08; First posted 2014-01-14 (Estimated); Last update posted 2017-04-06 (Actual); Status verified 2017-04

CONDITIONS: Uterine Cervical Cancer
Keywords: Locally advanced cervical cancer; Concurrent chemoradiation; Adjuvant chemotherapy
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Brachytherapy; Cisplatin; Pharmaceutical Preparations; Paclitaxel; Carboplatin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Concurrent chemoradiation (Active Comparator): Radiation: Radiation Therapy
  * External beam pelvic radiotherapy (45-50.4 Gy in 1.8 Gy fractions) delivered by Linear accelerator machine
  * Vaginal brachytherapy for 4-5 fractions
  Chemotherapy: Cisplatin
  - Cisplatin 40 mg/m2 i.v., q wk, 6 cycles during radiotherapy
  Interventions: Radiation: Pelvic radiation; Drug: Cisplatin
- Concurretn chemoradiation plus adjuvant chemotherapy (Experimental): Radiation: Radiation Therapy
  * External beam pelvic radiotherapy (45-50.4 Gy in 1.8 Gy fractions) delivered by Linear accelerator machine
  * Vaginal brachytherapy for 4-5 fractions
  Chemotherapy: Cisplatin, paclitaxel, carboplatin
  * Cisplatin 40 mg/m2 i.v., q wk, 6 cycles during radiotherapy
  * Paclitaxel 175 mg/m2 i.v. q 4 wks, 3 cycles starting 4 week after completion of CCRT
  * Carboplatin AUC 5 i.v. q 4 wks, 3 cycles given together with paclitaxel
  Interventions: Radiation: Pelvic radiation; Drug: Cisplatin; Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Radiation: Pelvic radiation — Radiation:
  * Pelvic radiation 1.8 Gy/ day, 5 days/ week, 6 weeks
  * Brachytherapy 30-35 Gy for 4-5 times
  Other Names: External beam pelvic radiation therapy and brachytherapy
Drug: Cisplatin — Cisplatin 40 mg/m2 i.v.
  Other Names: Drugs:; - Cisplatin; - Kemoplat®; - Platin®
Drug: Paclitaxel — Paclitaxel 175 mg m2 i.v.
  Other Names: - Intaxel®; - Anzatax®
  Arms: Concurretn chemoradiation plus adjuvant chemotherapy
Drug: Carboplatin — Carboplatin AUC 5 i.v.
  Other Names: - Carboplatin®; - Kemocarb®
  Arms: Concurretn chemoradiation plus adjuvant chemotherapy

SUMMARY:
Data of survival benefit from adjuvant chemotherapy (ACT) after concurrent chemoradiation (CCRT) for locally advanced cervical cancer (LACC) are still limited and inconsistent. We will investigate if ACT has survival benefit over CCRT alone.

DETAILED DESCRIPTION:
Concurrent chemoradiation (CCRT) is the standard treatment for cervical cancer of FIGO stage IIB-IVA or so called locally advanced cervical cancer (LACC). However, failure rate after treatment is still as high as 30% to 40%.

This is a multi-center randomized controlled trial which evaluates whether adjuvant chemotherapy (ACT) after CCRT will improve treatment outcome comparing to CCRT alone.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years
* Cervical cancer FIGO stage IIB-IVA
* Histopathology of squamous cell carcinoma, adenocarcinoma, or adenosquamous cell carcinoma
* ECOG performance status 0-2
* No history of other cancer except basal cell carcinoma
* Adequate bone marrow function (WBC > or = 3,000/mm3, granulocytes > or = 1,500/mm3, platelet count > or = 100,000/mm3)
* Bilirubin < 1.5 folds, SGOT/ SGPT < 1.5 folds of normal limit, creatinine clearance > or = 40 mg/dl
* Consent to participate

Exclusion Criteria:

* Para-aortic lymph node enlargement > 1 cm or suspicious for cancer metastasis from CT or MRI
* Adnexal mass from physical examination or imaging study
* Chronic illnesses e.g. renal failure/ impairment, peripheral or central neuropathy, uncontrolled diabetes mellitus, or HIV infection.
* Pregnancy or lactation

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2014-01; Primary Completion 2018-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 3 years
  3-year progression free survival

SECONDARY OUTCOMES:
Overall survival | 3 years
  3-year overall survival

OTHER OUTCOMES:
Response rate | 4 months after completion of CCRT
  Response rate will be assessed at 4 months after completion of CCRT (expected to be at 4 months after CCRT in the control arm or at 1 month after completion of adjuvant chemotherapy in the study arm)
Cost-utility analysis | Cost of treatment and quality of life will be assessed at baseline, completion of CCRT, q month for 3 months after CCRT, after each cycle of ACT, 2 years after completion of treatment, and when there are tumor persistence, progression or recurrence
  Cost and quality of life
Adverse event | up to 6 months after treatment
  Adverse events occurred during and after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Siriwan Tangjitgamol, MD, Principal Investigator — Navamindradhiraj University; Vichan Lordvithaya, MD, Principal Investigator — Chiang Mai University
Locations (11):
- Thailand (11):
  - Bhumibol Adulyadej Hospital, Bangkok, Bangkok
  - Department of Obstetrics and Gynecology, Department of Radiology, Epidemiology Unit, Navamindradhiraj University, Bangkok, Bangkok
  - Health Intervention and Technology Assessment Program, Bangkok, Bangkok
  - Chonburi Cancer Hospital, Chon Buri, Changwat Chon Buri
  - Lampang Cancer Hospital, Lampang, Changwat Lampang
  - Lopburi Cancer Hospital, Lopburi, Changwat Lop Buri
  - Ratchaburi Hospital, Muang, Changwat Ratchaburi
  - Department of Obstetrics and Gynecology, Department of Radiology, Prince of Songkla University, Songkhla, Changwat Songkhla
  - Department of Radiology, Department of Obstetrics and Gynecology, Chiang Mai University, Chiang Mai, Chiang Mai
  - Ubonratchathani Cancer Hospital, Ubonratchathani, Ubonratchathani
  - Udonthani Cancer Hopital, Udon Thani, Udonthani

REFERENCES:
- [Derived] Tangjitgamol S, Tharavichitkul E, Tovanabutra C, Rongsriyam K, Asakij T, Paengchit K, Sukhaboon J, Penpattanagul S, Kridakara A, Hanprasertpong J, Chomprasert K, Wanglikitkoon S, Atjimakul T, Pariyawateekul P, Katanyoo K, Tanprasert P, Janweerachai W, Sangthawan D, Khunnarong J, Chottetanaprasith T, Supawattanabodee B, Lertsanguansinchai P, Srisomboon J, Isaranuwatchai W, Lorvidhaya V. A randomized controlled trial comparing concurrent chemoradiation versus concurrent chemoradiation followed by adjuvant chemotherapy in locally advanced cervical cancer patients: ACTLACC trial. J Gynecol Oncol. 2019 Jul;30(4):e82. doi: 10.3802/jgo.2019.30.e82. Epub 2019 Apr 10. PMID 31074236